CLINICAL TRIAL: NCT02573363
Title: Phase I Investigator Sponsored Study to Assess the Tolerability and Efficacy of Selinexor in Combination With High Dose Cytarabine (HiDAC) and Mitoxantrone Chemotherapy for Remission Induction in Acute Myelogenous Leukemia (AML)
Brief Title: Selinexor With Combination Chemotherapy in Treating Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB15-0412; NCI-2015-01647 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB15-0412 (Other: University of Chicago Comprehensive Cancer Center); P30CA014599 (NIH)
Record Dates: First submitted 2015-10-05; First posted 2015-10-09 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Mitoxantrone; selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- selinexor, cytarabine, and mitoxantrone (Experimental): INDUCTION CHEMOTHERAPY: Patients receive high-dose cytarabine and mitoxantrone hydrochloride per standard of care on days 1 and 5, and selinexor PO on days 2, 4, 9, and 11.
  CONSOLIDATION CHEMOTHERAPY: Patients receive high-dose cytarabine per standard of care on days 1, 3, and 5, and selinexor PO on days 2, 4, 9, and 11. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE CHEMOTHERAPY: Patients achieving at least stable disease after consolidation chemotherapy may receive selinexor PO on days 1, 8, 15, and 22 at the discretion of principal investigator.
  Interventions: Drug: Cytarabine; Drug: Mitoxantrone Hydrochloride; Drug: Selinexor

INTERVENTIONS:
Drug: Cytarabine — Given per standard of care
  Other Names: Ara-C
Drug: Mitoxantrone Hydrochloride — Given per standard of care
  Other Names: Mitroxone
Drug: Selinexor — Given PO
  Other Names: KPT-330

SUMMARY:
This phase I trial studies the side effects and the best dose of selinexor when give together with standard chemotherapy, high dose cytarabine and mitoxantrone hydrochloride, in treating patients with acute myeloid leukemia. Selinexor may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cytarabine and mitoxantrone hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving selinexor together with standard chemotherapy may be a better treatment for patients with acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Signed, written informed consent in accordance with federal, local, and institutional guidelines
* Patients with newly diagnosed or relapsed/refractory AML, except acute promyelocytic leukemia (APL), requiring intensive induction chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Creatinine clearance > 30 cc/min calculated using the Cockcroft and Gault (1976) formula or measured
* Total bilirubin =< 2 mg/dl unless high indirect bilirubin is due to a congenital disorder
* Transaminases (aspartate aminotransferase [AST] or alanine aminotransferase [ALT]) =< 3.0 x upper limit of normal (ULN) unless due to leukemia infiltration
* Prothrombin time (PT) and partial thromboplastin time (PTT) =< 2 x ULN
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures
* It is important patients understand the need to use birth control while on this study; female patients of child-bearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test at screening (< 3 days prior to first dose), male patients with partners of childbearing potential must agree to use effective contraception during the study period and a period of 3 months after the last dose of study drug; for both male and female patients, effective methods of contraception must be used throughout the study and for three months following the last dose

Exclusion Criteria:

* Treatment with any investigational agent within two weeks prior to first dose in this study; hydroxyurea is allowed to control the AML prior to treatment on the study
* AML central nervous system (CNS) involvement
* Major surgery within 2 weeks of first dose of study drug; patients must have recovered from the effects of any surgery performed greater than 2 weeks previously
* Patient has a concurrent advantage active malignancy under treatment
* Unstable cardiovascular function:

  * Symptomatic ischemia, or
  * Uncontrolled clinically significant conduction abnormalities (i.e., ventricular tachycardia on antiarrhythmic agents are excluded; 1st degree atrioventricular [AV] block or asymptomatic left anterior fascicular block/right bundle branch block [left anterior fascicular block (LAFB)/right bundle branch block (RBBB)] will not be excluded), or
  * Congestive heart failure (CHF) New York Heart Association (NYHA) class >= 3, or
  * Myocardial infarction (MI) within 3 months
* Uncontrolled infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to first dose; infections controlled on concurrent anti-microbial agents are acceptable, and anti-microbial prophylaxis per institutional guidelines is acceptable
* Known active hepatitis B virus (HBV) or C virus (HCV) infection; or known to be positive for HCV ribonucleic acid (RNA) or HBsAg (HBV surface antigen)
* Known human immunodeficiency virus (HIV) infection
* Any medical condition which, in the investigator's opinion, could compromise the patient's safety
* Patients unable to swallow tablets or patients with malabsorption syndrome, or any other disease significantly affecting gastrointestinal function
* Seizure or cerebrovascular accident (CVA) in the last year

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-10-07 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2019-05-03 (Actual)

PRIMARY OUTCOMES:
MTD of selinexor based on the dose-limiting toxicity graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 | 56 days

SECONDARY OUTCOMES:
Allo-SCT success rate | After completion of induction therapy (6 months to a year)
Incidence of adverse events graded according to NCI CTCAE version 4.03 | Up to 30 days post-treatment
Incidence of non-relapse mortality | Up to 1 year
Overall survival (OS) rates | Date induction chemotherapy to the date of disease relapse or death, assessed up to 1 year
  The median duration of OS will be estimated based on the 50th percentile of the Kaplan-Meier distribution; additional summary statistics will be presented, including the 25th and 75th percentiles, 95% CIs on the median and other percentiles, and proportion of censored data. Kaplan-Meier survival rates will also be calculated.
Progression-free survival (PFS) rates | Date induction chemotherapy to the date of disease relapse or death, assessed up to 1 year
  PFS will be estimated based on the 50th percentile of the Kaplan-Meier distribution; additional summary statistics will be presented, including the 25th and 75th percentiles, 95% confidence intervals (CIs) on the median and other percentiles, and proportion of censored data. Kaplan-Meier survival rates will also be calculated.

OTHER OUTCOMES:
MRD status as measured by WT1 transcript levels using quantitative real time-PCR | Up to 1 year
  Cox models may be used to determine MRD status during the treatment course.

CONTACTS AND LOCATIONS:
Overall Officials: Hongtao Liu, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Wang AY, Weiner H, Green M, Chang H, Fulton N, Larson RA, Odenike O, Artz AS, Bishop MR, Godley LA, Thirman MJ, Kosuri S, Churpek JE, Curran E, Pettit K, Stock W, Liu H. A phase I study of selinexor in combination with high-dose cytarabine and mitoxantrone for remission induction in patients with acute myeloid leukemia. J Hematol Oncol. 2018 Jan 5;11(1):4. doi: 10.1186/s13045-017-0550-8. PMID 29304833